CLINICAL TRIAL: NCT00357669
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy and Safety of Brivaracetam Used as Adjunctive Treatment for 12 Weeks in Adolescent and Adult Patients (≥16 Years) With Genetically Ascertained Unverricht-Lundborg Disease
Brief Title: Brivaracetam as add-on Treatment of Unverricht-Lundborg Disease in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01187; 2006-000169-12 (EudraCT Number)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Unverricht-Lundborg Disease
Keywords: Unverricht-Lundborg disease; Baltic myoclonus; progressive myoclonic epilepsies; myoclonus; brivaracetam
MeSH Terms: conditions — Unverricht-Lundborg Syndrome; Myoclonic Epilepsies, Progressive; Myoclonus | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Brivaracetam 50 mg/day (Experimental): BRV 50 mg/day
  Interventions: Drug: Brivaracetam 25 mg; Drug: Brivaracetam 50 mg
- Brivaracetam 150 mg/day (Experimental): BRV 150 mg/day
  Interventions: Drug: Brivaracetam 25 mg; Drug: Brivaracetam 50 mg

INTERVENTIONS:
Drug: Brivaracetam 25 mg — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 25 mg
  * Route of Administration: Oral use
  Other Names: ucb34714
  Arms: Brivaracetam 150 mg/day; Brivaracetam 50 mg/day
Drug: Brivaracetam 50 mg — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Other Names: ucb34714
  Arms: Brivaracetam 150 mg/day; Brivaracetam 50 mg/day
Other: Placebo — * Active Substance: Placebo Pharmaceutical Form: Tablet
  * Concentration: 25 mg and 50 mg
  * Route of Administration: Oral use
  Arms: Placebo

SUMMARY:
The study will compare the efficacy and safety of brivaracetam with placebo in patients with Unverricht-Lundborg disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed Unverricht-Lundborg disease (ULD) ascertained by appropriate genetic testing for a homozygous or compound heterozygous mutation in the Cystatin B (CSTB) gene
* Subjects with moderate to severe myoclonus documented by an Action Myoclonus sum score of ≥ 30 (evaluation by investigator)
* Subjects currently being or having been treated with clonazepam up to the maximum recommended daily dose of 20 mg or up to their individual optimal dose as assessed by the investigator
* Subjects currently being or having been treated with valproate up to the maximum recommended daily dose 60 mg/kg or serum levels of 100 mcg/ml or up to their individual optimal dose as specified by the investigator

Exclusion Criteria:

* Subjects currently on felbamate or having been on felbamate within less than 18 months prior to Visit 1
* Subjects currently treated with phenytoin or having been on phenytoin in the last month prior to Visit 1
* Subjects currently on vigabatrine. Subjects having been on vigabatrine if no visual fields examination report available including standard static (Humphrey or Octopus) or cinetic perimetry (Goldman)
* Subject taking any drug with possible central nervous system (CNS) effects
* Subjects taking any drug that may significantly influence the metabolism of BRV (CYP2C or CYP3A potent inducers/inhibitors)
* Known clinically significant acute or chronic illness or illness which may impair reliable participation in the trial, necessitate the use of medication not allowed by protocol or represent a safety risk in the Investigator's opinion
* Subjects with history of severe adverse hematological reaction to any drug
* Impaired hepatic function: ALAT/SGPT, ASAT/SGOT, alkaline phosphatase, GGT value of more than three times the upper limit of the reference range
* History of suicide attempt during the last 5 years
* Subject with suicidal ideations within the last year or at risk of suicide attempt unless cleared by written confirmation from a psychiatrist and approved by the UCB physician
* Ongoing psychiatric disorder other than mild controlled disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline on the Action Myoclonus score (Unified Myoclonus Rating Scale (UMRS) Section 4) at the end of the Treatment Period | End of treatment period (Week 14 or early discontinuation visit)

SECONDARY OUTCOMES:
Percent reduction from baseline on the functional disability score (UMRS Section 5) at the end of the Treatment Period | End of treatment period (week 14 or early discontinuation visit)
Percent reduction from baseline on the stimulus sensitivity score (UMRS Section 3) at the end of the Treatment Period | End of treatment period (week 14 or early discontinuation visit)
Percent reduction from baseline on the myoclonus patient questionnaire (UMRS Section 1) at the end of the Treatment Period | End of treatment period (week 14 or early discontinuation visit)
Global Evaluation Scale by Investigator (I-GES) at the end of the Treatment Period | End of treatment period (week 14 or early discontinuation visit)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (13):
- Finland (2):
  - Kuopio
  - Tampere
- France (2):
  - Marseille
  - Montpellier
- Italy (4):
  - Bologna
  - Messina
  - Milan
  - Napoli
- Netherlands (2):
  - Heemstede
  - Heeze
- Saint Pierre Cedex, Reunion
- Gothenburg, Sweden
- Tunis, Tunisia

REFERENCES:
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041
- [Derived] Kalviainen R, Genton P, Andermann E, Andermann F, Magaudda A, Frucht SJ, Schlit AF, Gerard D, de la Loge C, von Rosenstiel P. Brivaracetam in Unverricht-Lundborg disease (EPM1): Results from two randomized, double-blind, placebo-controlled studies. Epilepsia. 2016 Feb;57(2):210-21. doi: 10.1111/epi.13275. Epub 2015 Dec 15. PMID 26666500